CLINICAL TRIAL: NCT00928694
Title: An Open-Label, Randomized, 2-Period, Crossover Study to Determine Definitive Bioequivalence After Administration of Single 160 mg Doses of the U.S. and UK Formulations of Fenofibrate in Healthy Adult Subjects
Brief Title: Fenofibrate Bioequivalence Study (0767-031)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0767-031; MK0767-031; 2009_606
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Results first posted 2009-12-11 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Fenofibrate

ARMS (2):
- 1 (Active Comparator): Fenofibrate U.S. Formulation
  Interventions: Drug: fenofibrate (U.S. formulation)
- 2 (Active Comparator): Fenofibrate UK Formulation
  Interventions: Drug: fenofibrate (UK formulation)

INTERVENTIONS:
Drug: fenofibrate (U.S. formulation) — Single dose of 160 mg fenofibrate U.S. formulation (Tricor®) in one of two treatment periods.
  Other Names: Tricor®
  Arms: 1
Drug: fenofibrate (UK formulation) — Single dose of 160 mg fenofibrate UK formulation (Supralip®) in one of two treatment periods.
  Other Names: Supralip®
  Arms: 2

SUMMARY:
This study will determine definitive bioequivalence of the United States (U.S.) and United Kingdom (UK) formulations of fenofibrate following administration of single doses in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health
* Subject is willing to follow all study guidelines

Exclusion Criteria:

* Subject has uncontrolled high blood pressure, impaired glucose tolerance, diabetes, or other major diseases or chronic conditions that would confound the results of the study or make participation unsafe
* Female subject is receiving oral contraceptives or hormone replacement therapy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2003-02; Primary Completion 2003-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- TRICOR™ First, Then SUPRALIP™: U.S. formulation (TRICOR™) 160 mg tablet/ UK formulation (SUPRALIP™) 160 mg tablet
- SUPRALIP™ First, Then TRICOR™: UK formulation (SUPRALIP™) 160 mg tablet / U.S. formulation (TRICOR™) 160 mg tablet
Period: First Intervention
Arm/Group | TRICOR™ First, Then SUPRALIP™ | SUPRALIP™ First, Then TRICOR™
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | TRICOR™ First, Then SUPRALIP™ | SUPRALIP™ First, Then TRICOR™
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: years] | 36.7 [23 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Height [Mean (Full Range); unit: Centimeters] | 169.64 [154.94 to 187.96]
Weight [Mean (Full Range); unit: Kilograms] | 73.94 [51.71 to 93.90]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC(0 to Infinity)) of Fenofibric Acid
Time Frame: Predose and up to 168 hours postdose
Population: Healthy Male and Female subjects Aged 18 to 45
Measure: Least Squares Mean (Standard Deviation); unit: μg·hr/mL
Groups:
- U.S. Formulation (TRICOR™): U.S. Formulation: single oral 160 mg dose of the U.S. formulation of fenofibrate with food.
- UK Formulation (SUPRALIP™): UK Formulation: single oral 160 mg dose of the UK formulation of fenofibrate with food.
Arm/Group | U.S. Formulation (TRICOR™) | UK Formulation (SUPRALIP™)
Number analyzed (Participants) | 14 | 14
μg·hr/mL | 116 (35.1) | 121 (36.4)
Statistical Analysis 1: Comparison: U.S. Formulation (TRICOR™) vs UK Formulation (SUPRALIP™); Test type: Non-Inferiority or Equivalence — Bioequivalence bounds = (0.80, 1.25) Study Primary Hypothesis: Single 160 mg doses of the U.S. and UK formulations of fenofibrate following consumption of a standard breakfast are bioequivalent (the true geometric mean ratios (GMRs) [U.S./UK] for the AUC(0 to infinity) and maximum plasma concentration (Cmax) of fenofibric acid after administration of the U.S. and UK formulations of fenofibrate with food are contained in the interval [0.80, 1.25]); Geometric Mean Ratio = 0.96, 90% CI [0.90 to 1.02]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Fenofibric Acid
Time Frame: Predose and up to 168 hours postdose
Population: Healthy Male and Female subjects Aged 18 to 45
Measure: Least Squares Mean (Standard Deviation); unit: μg/mL
Arm/Group | U.S. Formulation (TRICOR™) | UK Formulation (SUPRALIP™)
Number analyzed (Participants) | 14 | 14
μg/mL | 6.35 (1.61) | 6.48 (1.80)
Statistical Analysis 1: Comparison: U.S. Formulation (TRICOR™) vs UK Formulation (SUPRALIP™); Test type: Non-Inferiority or Equivalence — Bioequivalence bounds = (0.80, 1.25) Study Primary Hypothesis: Single 160 mg doses of the U.S. and UK formulations of fenofibrate following consumption of a standard breakfast are bioequivalent (the true GMRs [U.S./UK] for the AUC(0 to infinity) and Cmax of fenofibric acid after administration of the U.S. and UK formulations of fenofibrate with food are contained in the interval [0.80, 1.25]); Geometric Mean Ratio = 0.98, 90% CI [0.90 to 1.06]

ADVERSE EVENTS:
Groups:
- Tricor™: U.S. formulation (TRICOR™) 160 mg tablet
- Supralip™: UK formulation (SUPRALIP™) 160 mg tablet
Arm/Group | Tricor™ | Supralip™
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tricor™ (N=14) | Supralip™ (N=14)
Loose Stools (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.